CLINICAL TRIAL: NCT05507528
Title: EVALUATION OF THE SAFETY AND EFFICACY OF REBORN LED SYSTEM FOR NON-INVASIVE LIPOLYSIS TREATMENT
Brief Title: Evaluation of the Safety and Efficacy of REBORN System for Lipolysis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lightfective Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-LF-01
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: LIPOLYSIS

STUDY DESIGN:
Intervention Model Description: open label, prospective, single arm, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Reborn treatment group (Experimental): The Lightfective ReBorn System is a Diode Light Emitting Diode (LED) System, Fat reduction treatments with the ReBorn LED System visit - include the treatment procedure
  Interventions: Device: reborn treatment

INTERVENTIONS:
Device: reborn treatment — Fat reduction treatments with the ReBorn LED System visit - include the treatment procedure

SUMMARY:
The Lightfective ReBorn System is intended for non-invasive lipolysis of the flanks in individuals with a Body Mass Index (BMI) of 30 or less. The device is intended to affect the appearance of visible fat bulges in the flanks.

DETAILED DESCRIPTION:
Body countering and fat reduction treatment are considered to be one of the most popular aesthetic procedures. The Lightfective' ReBorn LED System provides non-invasive fat reduction treatment.

The primary efficacy objective is to demonstrate fat reduction in the treated area after treatment with the ReBorn LED system.

study population, Healthy subjects who seek for fat reduction treatments in the flanks area.

Each subject will undergo 2 treatment visits (one month apart) and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 22 years of age.
2. Subject has clearly visible fat on the flanks area.
3. Subject has not experienced weight change exceeding 4.5kg in the preceding month.
4. Subject agrees to maintain their weight (i.e., within 2.25kg) by not making any major changes in their diet or lifestyle during the course of the study.
5. Subject is willing and able to comply with protocol requirements and all study visits
6. Subject has provided a written informed consent

Exclusion Criteria:

1. Subject underwent a prior surgical procedure(s) in the area of intended treatment within the past 6 months.
2. Subject underwent a prior invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment within the past year.
3. Subject underwent a prior non-invasive fat reduction procedure in the area of intended treatment within the past 6 months.
4. Subject has a known history of subcutaneous injections into the area of intended treatment (e.g., clexane, insulin) within the past month.
5. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
6. Subject has a known history of Reynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
7. Subject has a history of bleeding disorder, or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
8. Subject body mass index (BMI) exceeds 30. BMI is defined as weight in kg divided by the square of the height in cm.
9. Subject is taking or has taken diet pills or supplements within the past month.
10. Subject has any dermatological conditions or scars in the location of the treatment sites that may interfere with the treatment or evaluation.
11. Subject is pregnant or intending to become pregnant in the next 6 months.
12. Subject is lactating or has been lactating in the past 6 months.
13. Subject is unable or unwilling to comply with the study requirements.
14. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
15. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.
16. Subject is currently taking weight reduction medications (e.g., Saxenda).
17. Subject is currently taking GLP-1 receptor agonist medications (e.g., Victoza).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Fat reduction | 20 weeks
  to demonstrate fat reduction in the treated area after treatment with the ReBorn LED system.
Blinded reviewers evaluation | 20 weeks
  subject's pre and post-treatment photographs will be presented in randomized order to blinded reviewers for evaluation.
  Subject is considered "success" if at least two out of the three evaluators correctly identify photographs order.

SECONDARY OUTCOMES:
safety evaluation | 20 weeks
  The safety of the ReBorn LED System will be demonstrated by serious adverse event during the study.

CONTACTS AND LOCATIONS:
Locations (3):
- Tennessee Clinical Research Center, Tennessee City, Tennessee, United States
- Israel (2):
  - Herzelia Medical Center - Tal Nachliely clinic, Kiryat Bialik
  - rabin medical center - campus Hasharon, Petah Tikva

IPD SHARING:
Plan to Share IPD: No